CLINICAL TRIAL: NCT01831830
Title: Evaluation of the Veterans' In-home Programs for Veterans With TBI and Families
Brief Title: Evaluation of the Veterans' In-home Program
Acronym: VIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporal Michael J. Crescenz VA Medical Center (U.S. Federal Agency)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Laraine Winter, Research Psychologist, Corporal Michael J. Crescenz VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01308; 1R21HD068857-01 (NIH)
Record Dates: First submitted 2013-04-11; First posted 2013-04-15 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; occupational therapy; family
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- control condition (No Intervention): The control group receives two attention-control calls.
- The Veterans' in-home program (Experimental): The VIP intervention consists of 8 sessions (up to 6 in the home and 2 phone calls) from an occupational therapist. This is delivered to Veterans and their family members.
  Interventions: Behavioral: The Veterans' In-home Program

INTERVENTIONS:
Behavioral: The Veterans' In-home Program — VIP realigns environmental demands to match Veterans' abilities through the modification of home environments, development of meaningful activities tailored to Veterans' strengths, training in the use of emotion-regulation strategies to address behavioral/interpersonal difficulties, and training in the use of cognitive strategies to compensate for cognitive impairments. In its family focus, VIP provides family members with education and training to understand and manage the Veterans' limitations.
  Arms: The Veterans' in-home program

SUMMARY:
The primary objective of this study is to evaluate the preliminary effectiveness and acceptability of an innovative in-home nonpharmacological intervention, the Veterans' In-home Program (VIP), for Veterans with mild to moderate traumatic brain injury (TBI) and their families. VIP is designed to promote community reintegration, improve quality of life, and support functioning by realigning environmental demands to match the Veteran's abilities.

DETAILED DESCRIPTION:
Research Design: Using a 2-group randomized control trial, the investigators will evaluate the intervention in comparison to usual care. Usual care is traditional clinic-based care, which will be enhanced by 2 phone calls to provide an attention control condition.

Methodology: Participants will be 100 Veterans diagnosed with mild to moderate TBI who are followed by the Philadelphia VA Medical Center (PVAMC) Polytrauma Service and a family member (100) of each Veteran. All Veterans will have a family member or partner living with them who is willing to participate in the study. The intervention and study interviews will occur in Veterans' homes. Qualitative phone interviews with a subset of the sample who received the intervention will be conducted at PVAMC.

Primary study outcomes for the Veterans will be physical, cognitive, and emotional/interpersonal functioning and community reintegration, measured by standardized instruments at baseline and follow-up at 3 to 4 months. Study outcomes for family members will be mood and dimensions of well-being, measured by standardized instruments at baseline and follow-up at 3 to 4 months. Acceptability of the intervention for Veterans and family members will be measured through Project Evaluations, administered at follow-up with both groups. In addition, qualitative phone interviews will be conducted with a subset of Veterans and family members who received VIP to evaluate VIP's acceptability and to enhance understanding of the impact of VIP from the perspective of those experiencing it.

Based on a person-environment fit framework, the VIP intervention consists of 8 sessions (up to 6 in the home and 2 telephone contacts) delivered by occupational therapists over a 3 month period to Veterans and family members. VIP realigns environmental demands to match Veterans' abilities through the modification of home environments, development of meaningful activities tailored to Veterans' strengths, training in the use of emotion-regulation strategies to address behavioral/interpersonal difficulties, and training in the use of cognitive strategies to compensate for cognitive impairments. In its family focus, VIP provides family members with education and training to understand and manage the Veterans' limitations.

Clinical relationships: VIP extends and adds value to traditional on-site clinical care by helping individuals with TBI and their families in the setting where most functional and behavioral problems emerge. As a skills-building intervention, VIP has the potential to enhance Veterans' abilities to function effectively in their home environments and to improve their quality of life and that of their families.

ELIGIBILITY:
Inclusion Criteria:

* patient with mild-moderate TBI followed by PVAMC Polytrauma Service
* English speaking
* a family member/partner living with or nearby who is willing to participate in the study

Exclusion Criteria:

* At high risk for violence
* currently receiving in-home service

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2011-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Preliminary effectiveness and acceptability for Veteran | 4 months
  Preliminary effectiveness includes Veterans' physical, cognitive, and emotional/interpersonal functioning and community reintegration. Acceptability is measured through project evaluations and qualitative interviews.

SECONDARY OUTCOMES:
Preliminary effectiveness and acceptability for family member | 4 months
  Preliminary effectiveness is measured through mood and dimensions of well-being. Acceptability is measured through project evaluations and qualitative interviews.

OTHER OUTCOMES:
Refinement of intervention procedures and assessment tools | 4 months
  The Delivery Assessments describe characteristics of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Laraine Winter, PhD, Principal Investigator — Philadelphia VA Medical Center, The Philadelphia Research & Education Foundation; Helene J Moriarty, PhD, RN, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center
Locations (1):
- Philadelphia VA Medical Center, Philadelphia, Pennsylvania, United States